CLINICAL TRIAL: NCT06524219
Title: A Prospective, Multi-center, Real-world Study on the Comparison of Different Nerve-sparing Techniques in Retzius-sparing Robot-assisted Radical Prostatectomy for Oncological Outcome and Functional Recovery.
Brief Title: Comparison of Nerve-sparing Techniques in Radical Prostatectomy for Oncological Outcome and Functional Recovery.
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-SR-394
Record Dates: First submitted 2024-07-17; First posted 2024-07-29 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- unilateral intrafascial resection: Subjects whose preoperative MRIs indicate the lesions are located in the peripheral zone of one side near the capsule, unable to be performed intrafascial resection, and no major lesion or only slight lesion in the peripheral zone of the other side, are going to be conducted unilateral intrafascial resection in Retzius-sparing robot-assisted radical prostatectomy.
  Interventions: Procedure: unilateral intrafascial resection
- bilateral intrafascial resection: Subjects who have low or median-risk tumors and no extracapsular extension for major lesion, are going to be conducted bilateral intrafascial resection in Retzius-sparing robot-assisted radical prostatectomy.
  Interventions: Procedure: bilateral intrafascial resection
- bilateral extrafascial resection: Subjects who have major lesion that is in the peripheral zone, MRIs that show that the lesion may invade or locate at the edge of the transitional zone, and Gleason score of 4+4 or greater, are going to be conducted bilateral intrafascial resection in Retzius-sparing robot-assisted radical prostatectomy.
  Interventions: Procedure: bilateral extrafascial resection

INTERVENTIONS:
Procedure: unilateral intrafascial resection — Conducting unilateral intrafascial resection in Retzius-sparing robot-assisted radical prostatectomy
  Groups: unilateral intrafascial resection
Procedure: bilateral intrafascial resection — Conducting bilateral intrafascial resection in Retzius-sparing robot-assisted radical prostatectomy
  Groups: bilateral intrafascial resection
Procedure: bilateral extrafascial resection — Conducting bilateral extrafascial resection in Retzius-sparing robot-assisted radical prostatectomy
  Groups: bilateral extrafascial resection

SUMMARY:
To evaluate the difference among three nerve-sparing techniques(unilateral intrafascial resection, bilateral intrafascial resection, bilateral extrafascial resection) of oncological outcome and functional recovery.

DETAILED DESCRIPTION:
Surgery is a common and effective treatment for localized prostate cancer. The main objective of surgical treatment is to remove the tumor completely in order to achieve the goal of cure. Intrafascial nerve-sparing radical prostatectomy is a radical resection of prostate cancer with minimal damage to the nerves and blood vessels.

There are nerves around the prostate that affect sexual function, and damage to these nerves can lead to complications like sexual dysfunction and incontinence. Therefore, how to completely remove the tumor, as far as possible to preserve these nerves, become an important issue in the surgical treatment.

This study is aim to evaluate the different among nerve-sparing strategies, including unilateral intrafascial resection, bilateral intrafascial resection and bilateral extrafascial resection, on oncological outcome and functional recovery, so as to provide clinical evidence for nerve-sparing surgery of prostate cancer via robot-assisted posterior approach.

ELIGIBILITY:
Inclusion Criteria:

* Men aged ≥18 years and ≤80 years;
* Histologically proven prostate adenocarcinoma with clinical stage < T3(no capsule break)
* Clinically localized prostate cancer in very low, low, or intermediate risk groups according to National Comprehensive Cancer Network(NCCN) guidelines (2019 v4) ;
* Eastern Cooperative Oncology Group(ECOG) score of 0 or 1;
* Life expectancy greater than 10 years;
* Patients who are willing to accept robot-assisted radical prostatectomy after informed existing treatment plan, must sign the informed consent form.

Exclusion Criteria:

* Surgeon thinks that the patient has an unresectable disease;
* patients who have already applied androgen deprivation therapy(ADT);
* Preoperative images suggest that the local lymph nodes were larger than 2 cm or suggest bone or distant metastasis;
* Any contraindication;
* Previous treatment of prostate cancer, including but not limited to surgery, hormone therapy, chemotherapy, radiotherapy, targeted therapy and immunotherapy;
* Patients with a history of transurethral resection or enucleation of the prostate;
* Severe systemic disease that may interfere with the data, assessment, or compliance;
* Patients who are participating in other clinical trials;
* Refusing to sign the informed consent
* Patients that are considered to be not suitable to be included by the researchers.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients with prostate cancer who are willing to accept nerve-sparing techniques in Retzius-sparing robot-assisted radical prostatectomy, age between 18 to 80.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
biochemical recurrence-free rates | 3 years
  the rate of patients who do not have biochemical recurrence
urinary control rate | day 0, 3 month, 6 month, 1 year
  the rate of patients who do not have incontinence
sexual function | 6 month, 1 year
  the rate of patients who do not lose sexual function

SECONDARY OUTCOMES:
perioperative complications | perioperation
  the complications that occur in perioperation
positive rate of incisal margin | day 0
  the rate of patients who have positive incisal margin after the operation
prostate cancer-specific survival | 3 years
  the survival for prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Pengfei Shao, chief physician, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University